CLINICAL TRIAL: NCT03710226
Title: Is There an Association Between Platelet Indices and Recurrent Miscarriage?
Brief Title: Use of Platelet Indices for Prediction of Recurrent Miscarriage
Status: Completed | Type: Observational
Sponsor: Rania Hassan Mostafa (Other)
Responsible Party: Sponsor-Investigator, Rania Hassan Mostafa, Lecturer, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Other Study IDs: FMASU 1210/2018
Record Dates: First submitted 2018-10-13; First posted 2018-10-18 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Recurrent Miscarriage
Keywords: mean platelet volume; plateletcrit; platelet distribution width
MeSH Terms: conditions — Abortion, Habitual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: women with recurrent miscarriage (two or more consecutive miscarriages)
- controls: women without recurrent miscarriage and delivered at least once before

SUMMARY:
Platelet indices might be a marker for platelet activation, and thus could predict thrombosis. This might be the cause in some cases of recurrent miscarriage. This study aims to evaluate the use of platelet indices -as a simple test- to predict recurrent miscarriage.

DETAILED DESCRIPTION:
* Study population:
* Sample size: This study will be conducted on (70) women attending outpatient clinic divided into two groups:

  * 1st Group (35): women with history of recurrent miscarriage (two or more consecutive miscarriages)
  * 2nd Group (35): women without history of recurrent miscarriage and delivered at least once before.
* Sample size justification: The means of the platelet indices were used to calculate the sample size. Group sample sizes of 35 per group achieve 80% power to reject the null hypothesis of zero effect size when the population effect size is 0.70 (moderate to large) and the significance level (alpha) is 0.050 using a two-sided two-sample equal-variance t-test. (Machin et al., 1997)
* Methods:
* Enrollment: Women will be enrolled from the outpatient clinic and recurrent pregnancy loss outpatient clinic in Ain shams maternity hospital. 70 women will be enrolled from each clinic.
* Informed Consent: All participants will give their informed consent prior to enrollment
* Detailed history and general examination: To exclude obese women (BMI >30%), women with known uterine anomalies, endocrinological diseases or immunological disorders and women on anticoagulants or antiplatelet medications
* Transvaginal ultrasound: to exclude any uterine anomalies.
* Laboratory blood sampling: For testing of (TSH, HbA1C, Anticardiolipin antibody (IgG, IgM), lupus anticoagulant antibodies and Anti-β2 glycoprotein I ) in women with history of recurrent miscarriage and excluded if positive.

  * All other enrolled women will be tested by CBC by XN-1000(SA-01) machine.
  * The blood sample will be preserved by EDTA and will be processed within maximum 2 hours..
* Data collection & recording: Data of each patient will be recorded in a Case Record Form (CRF)
* Statistics:

Descriptive statistics for measured variables will be expressed as range, mean and standard deviation (for metric data); range, median and interquartile range (for discrete data); and number and proportions (for categorical data the platelet indices in each clinic will be compared using the t-test A P-value of 0.05 or less will be considered statistically significant.

• Ethical considerations:

1. Informed Consent Forms: Before being admitted to the study, the patient must consent to participate after the nature, scope, and steps of the study have been explained in a form understandable to her.

2- Confidentiality: Only the patient number and patient initials will be recorded in the CRF. The investigator will maintain a personal patient identification list (patient numbers with the corresponding patient names) to enable records to be identified.

3- Protocol approval: Before the beginning of the study and in accordance with the local regulation followed, the protocol and all corresponding documents will be declared for ethical and research approval by the council of obstetrics and gynaecology department, Ain Shams University; according to the WMA Declaration of Helsinki

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-49 years.
2. Women with history of recurrent miscarriage(two or more consecutive miscarriages)
3. Women with history of previous deliveries.

Exclusion Criteria:

1. Pregnant women
2. Women with medical disease (e.g. DM, thyroid disorders, hypertension, systemic lupus erythematosus, antiphospholipid antibody syndrome).
3. Women with known uterine anomalies.
4. Obesity (BMI >30%).
5. Women on anticoagulant medications or antiplatelet medications.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: women attending recurrent pregnancy loss clinic in Ain Shams University Maternity Hospital
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Mean Platelet Volume (MPV) | 1 day (measured once the participant is enrolled in the study & meets the eligibility criteria)
  it's a measure of the average size of the platelet, expressed in femtolitre (fL)
plateletcrit (PCT) | 1 day (measured once the participant is enrolled in the study & meets the eligibility criteria)
  it's a measure of total platelet mass, expressed in percentage (%).
Platelet Distribution Width (PDW) | 1 day (measured once the participant is enrolled in the study & meets the eligibility criteria)
  it's a measure that reflects variation of platelet size distribution, expressed in femtolitre (fL)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed k Makled, Phd, Study Chair — Professor; Wessam M Abuelghar, Phd, Study Director — Assistant professor
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt